CLINICAL TRIAL: NCT01707979
Title: NIR (Near Infrared)- Spectroscopy and Multifrequent Impedance Spectroscopy on the Skin to Detection of Sensory and Autonomic Neuropathy Among Patients With Type 1 Diabetes
Brief Title: NIR- and Multifrequent Impedance Spectroscopy on the Skin in Type 1 Diabetes
Acronym: NIR
Status: Completed | Type: Observational
Sponsor: Lise Tarnow (Other)
Responsible Party: Sponsor-Investigator, Lise Tarnow, Professor, Chief Physician, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Other Study IDs: NIR
Record Dates: First submitted 2012-09-25; First posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Diabetic Neuropathy
Keywords: Near infrared light; Diabetic neuropathy; Sensory neuropathy; Autonomic neuropathy; Vagus; Sudomotor function; Monofilament; Impedance
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Diabetic neuropathy: Male participants, type1 diabetic with diabetic neuropathy
- Diabetes without neuropathy: Male participants, type1 diabetic without diabetic neuropathy
- Non diabetic control: Male participants, control group non diabetic

SUMMARY:
The aim of the study is to examine the suitability to detect diabetic neuropathy using NIR and impedance.

DETAILED DESCRIPTION:
The aim of the study is to examine how suitable a hand-held measuring probe (DDD-probe) using NIR (near infrared light) as well as impedance (conductivity), is to detect early signs of diabetic neuropathy.

The DDD-probe is put directly on the skin and is measuring by the use of light and impedance.

ELIGIBILITY:
Inclusion Criteria:

* men with type 1 diabetes (WHO criteria)
* age 35-50 years
* duration of diabetes > 10 years

Exclusion Criteria:

* P-creatinine> 120 micromol/l
* other acute or chronic disease, or type of treatment that makes the patient unsuitable to participate, valuated by the investigator
* non intact skin on the measuring spots
* the patient is unable to understand the informed consent

Ages: 35 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Control group men without diabetes Type1 diabetic men without neuropathy complications Type 1 diabetic men with neuropathy complications
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
near infrared spectroscopy | one time
  Near infrared (NIR) is measured by spectroscopy on the skin using the DDD probe

CONTACTS AND LOCATIONS:
Overall Officials: Lise Tarnow, Professor, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark